CLINICAL TRIAL: NCT02429349
Title: Surgical Ovarian Preservation in Females Undergoing Chemo-Radiotherapy
Brief Title: Preservation of Ovarian Tissue and Chemo-Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-02542-FB
Record Dates: First submitted 2015-03-23; First posted 2015-04-29 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Endocrine Disorders of Female Reproductive System; Secondary Infertility; Infertility Involuntary
MeSH Terms: interventions — Surgical Procedures, Operative; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic Procedure (Experimental): Surgery - Unilateral surgical removal of ovary, freezing of tissue, post cancer cure autotransplant
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — Surgical Procedures- Unilateral oophorectomy will be performed by laparoscopy prior to undergoing chemo-radiation treatment as specified above. Subsequent ovarian cortex autotransplant will be performed by laparoscopy after the patients have been declared cured by their physicians.
  Other Names: surgical removal-ovary, freezing-tissue, autotransplant

SUMMARY:
The purpose of this study is to assess the results of ovarian tissue freezing, such as resumption or initiation of menses (menstruation: the discharge of blood and tissue from the uterus that happens about every 4 weeks in females who are not pregnant) and pregnancy, prior to starting chemotherapy or radiation treatment (commonly used for cancer treatment or for other conditions such as multiple sclerosis, psoriasis, rheumatoid arthritis). Females who are about to undergo chemotherapy or radiation therapy for cancer or these other medical conditions may stop having menses and may not be able to produce a biological child. Girls who have not achieved puberty and are exposed to chemotherapy (alkylating agents) or radiation treatment, the risk is up to 22-50%. In contrast, girls older than 10 years, or who have achieved puberty, experience acute ovarian failure in over 50% of the cases. By freezing and preserving ovarian tissue will help prevent these outcomes. In fact, when you are considered cured of your disease, you will have another surgical procedure where your own ovarian tissue will be transplanted back to you. This surgery will increase the possibility of resuming/initiating menses and the chance to have a pregnancy.

DETAILED DESCRIPTION:
At the present time, freezing of ovarian tissue is considered experimental and so thawing and future use of the tissue to initiate a pregnancy must be performed as part of a research program. With the patient's permission, a portion of her ovarian tissue will be frozen for her own use and a portion will be donated to a research pool.

Twenty subjects/year will be participating in this study.

Participation in this study will last until the patient's ovarian tissue is all used, or the patient decides to drop out of the study, or for the rest of her life. Freezing of ovarian tissue can be done only for research. Thawing and future use of the tissue to start a pregnancy must be done as part of a research program. After the age of 18, the patient will decide how and at what institution she wishes to use her own tissue in the future, for the purposes of becoming pregnant. The number of visits will be decided by the surgical procedure performed. The Investigators will contact the patient by phone, email, or mail until she has turned 18 years old, used her tissue or dropped out of the study (whichever comes first) to follow the patient's medical and fertility status over time and to ask questions about any future use of her frozen tissue and the possible results of the treatment. Depending on the patient's age at the time of enrollment, follow-up might be up to 30 years.

PURPOSE Primary objective: To assess resumption/initiation of menses after surgical ovarian preservation (ovarian tissue explant followed by freezing and autologous transplantation).

Secondary objective: To assess pre- and post-treatment production of various hormones, i.e., anti-mullerian hormone (AMH), insulin-like growth factor-1 (IGF-1), inhibin-B, follicle stimulating hormone (FSH), luteinizing hormone (LH), and estradiol, by serum and histological measurements.

Tertiary objective: To assess long-term sexual development, fertility competence, and lifespan of ovarian preservation via surgical autotransplant.

RATIONALE Chemotherapy treatment with alkylating agents and/or total body irradiation will prevent normal pubertal development of uterus, ovaries, and breasts because of primary ovarian insufficiency (POI). Explant and autologous transplantation of ovarian tissue will prevent ovarian insufficiency and allow normal sexual development through puberty and fertility competence.

RESEARCH DESIGN Prospective cohort study.

STUDY PROCEDURES Subject Recruitment and Screening- Subjects will be recruited by referral from the St. Jude Children's Research Hospital (SJCRH) and Methodist-Le Bonheur physicians to the Reproductive Medicine clinics held by Dr. Laura Detti. Patients will undergo an informed consent process in accordance with St. Jude Children's Research Hospital (SJCRH) and Methodist-Le Bonheur Institutional Review Boards.

Screening Visit- Complete medical history and physical exam; vital signs, height, and weight. Psychological Consult on impact of therapy.

Laboratory testing- Lab results for Estradiol, follicle stimulating hormone (FSH), luteinizing hormone (LH), Anti-Mullerian hormone (AMH), Inhibin B, will be obtained from the patients' clinical charts. In addition, Electrocardiogram (ECG) (12-lead); Bone age scan (if pre-pubertal), Pelvic ultrasound (transabdominal or transvaginal, depending on the patient's age) will be obtained from the patients' clinical charts. If a pelvic ultrasound has not been obtained prior to surgery, the procedure will be performed under anesthesia prior to the patient undergoing surgery for ovarian tissue harvesting).

Surgical Procedures- Unilateral oophorectomy will be performed by laparoscopy prior to undergoing chemo-radiation treatment as specified above. Subsequent ovarian cortex autotransplant will be performed by laparoscopy after the patients have been declared cured by their physicians.

Laparoscopic procedures- Upon general anesthesia is induced, attention will be turned to the patient's abdomen where 3-4 0.5 cm skin incisions will be performed (one in the umbilical fold and 2 lateral incisions; possibly, a 4th suprapubic incision). Disposable, bladed, trocars will be inserted in the abdominal cavity. The ovaries will be identified and a unilateral oophorectomy will be performed by retroperitoneal clamping/dissection of the infundibulo-pelvic and utero-ovarian ligaments.

A bipolar electrode will be used to assure accurate hemostasis and irrigation will be performed as needed. Upon retrieval of the trocars from the abdomen, the skin incisions will be reapproximated with 4-0 vycril sutures.

The second laparoscopic procedure will be done to perform autologous ovarian tissue transplant by suturing the thawed cortex fragments to the recipient ovary using 7-0 Prolene (Ethicon, Johnson and Johnson, USA), using the technique described by Silber et al. (Silber et al., 2005; Silber and Gosden, 2007) applied during laparotomy for transplantation.

As the transplanted tissue exhausts its function after the 1st autologous transplant, other laparoscopic procedures might become necessary over the years to transplant the rest of the cryopreserved tissue until no more tissue is available in the cryobank storage.

Freezing Procedure- The process of vitrification will be started in the Operating Room or in the lab within 120 minutes from collection of the sample and will be completed in the University of Tennessee Center for Reproductive Medicine laboratory. The tissue will be subdivided into numerous vials for individual storage/thawing. This will allow selective thawing for autotransplant over multiple procedures, if necessary.

Embryology laboratory procedures- The ovarian tissue that is stored for the patients will be used for autologous transplant. However, other techniques that are performed in the embryology laboratory may be available to the patients in the near future and might represent the best option for fertility preservation in patients with blood-borne cancers (i.e.: leukemia), in whom the risk of re-seeding cancer cells with tissue transplant is high.

Follow-Up Evaluation- Study treatment will include a post-operative visit and following scheduled follow-up visits for the patients' initial disease during which a complete physical exam and psychological evaluation will be conducted, and laboratory testing will be obtained for follicle stimulating hormone (FSH), luteinizing hormone (LH), anti-mullerian hormone (AMH), and Inhibin B.

Visits will be scheduled one month after explant and every 6-12 months until autotransplant of tissue and afterwards.

Laboratory testing, Electrocardiogram (ECG) (12-lead), Bone age, Pelvic ultrasound may be repeated yearly, as part of the patient's scheduled follow-ups. Bone age assessment will stop when a bone age of 18 years is achieved.

Patients who are going to develop ovarian insufficiency prior to or after puberty will undergo estrogen/progesterone therapy as per our institutional protocols.

Follow-up will continue until the patient stays enrolled in the study or until she reaches 40 years of age, or she goes in menopause and does not have, or does not desire, further tissue for transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Pre- and post-pubertal patients who are diagnosed with conditions that necessitate chemo- or radiotherapy and wish to preserve their ovarian function.

Exclusion criteria:

1. Patients with acute or chronic conditions that would preclude surgery. These include, but are not limited to, hyper- or hypo-coagulation disorders, lung conditions precluding mechanical ventilation, brain death.
2. Patients for whom the primary oncologist and/or pathologist discourage entering the protocol because of specific condition characteristics. These include, but are not limited to, cancers with high risk of ovarian metastasis such as leukemia and non-Hodgkin lymphoma.
3. Patients with known positive bone marrow for leukemia or solid tumor.
4. Patients whose tumor is in an organ that communicates with the peritoneum and peritoneal sampling at time of primary excision shows evidence of disease.
5. Patients older than 40 years of age.
6. Males.

Ages: 8 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05; Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Resumption of menses | Post-op, after initial explant surgery, & one month after, & every 6-12 months until autotransplant of tissue; through 40 yrs of age/menopause (or, pt.decision to stop earlier)
  Timing for resumption menses- patient report, physical evaluation at stated intervals.
Initiation of menses | Post-op, after initial explant surgery, & one month after, & every 6-12 months until autotransplant of tissue; through 40 yrs of age/menopause (or, pt.decision to stop earlier)
  Timing for initiation of menses- patient report, physical evaluation at stated intervals
Completion of puberty | Post-op, after initial explant surgery, & one month after, & every 6-12 months until autotransplant of tissue; through 40 yrs of age/menopause (or, pt.decision to stop earlier)
  Timing for completion of puberty - patient report, physical evaluation at stated intervals
Fertility | Post-op, after initial explant surgery, & one month after, & every 6-12 months until autotransplant of tissue; through 40 yrs of age/menopause (or, pt.decision to stop earlier)
  Timing for initiation of pregnancy - patient report, physical evaluation at stated intervals

SECONDARY OUTCOMES:
Physical UTERINE development | Follow-up at stated intervals, up to 30 years
  Physical assessment and pelvic ultrasound to evaluate uterine development before and after chemo- or radiotherapy treatment. Lifespan of transplanted cortex function (patient follow-up).
Physical OVARIAN development | Follow-up at stated intervals, up to 30 years
  Physical assessment and pelvic ultrasound to evaluate ovarian development before and after chemo- or radiotherapy treatment. Lifespan of transplanted cortex function (patient follow-up).

OTHER OUTCOMES:
Comparison of biochemical markers, i.e., Estradiol, FSH; LH, AMH; Inhibin B | Follow-up at stated intervals, up to 30 years
  Evaluation of biometry and of specific biochemical markers in the serum before and after chemo/radiation treatment and ovarian tissue explant, and in ovarian samples.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Detti, M.D., Principal Investigator — Associate Professor, UTennessee Health Science Center
Locations (7):
- United States (7):
  - Methodist/LeBonheur Hospital, Germantown, Tennessee
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Regional One Health Ob-Gyn Clinic, Memphis, Tennessee
  - Regional One Health, Regional Medical Center, Operating Room, Memphis, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee

REFERENCES:
- [Background] Meirow D, Lewis H, Nugent D, Epstein M. Subclinical depletion of primordial follicular reserve in mice treated with cyclophosphamide: clinical importance and proposed accurate investigative tool. Hum Reprod. 1999 Jul;14(7):1903-7. doi: 10.1093/humrep/14.7.1903. PMID 10402415
- [Background] Oktem O, Oktay K. A novel ovarian xenografting model to characterize the impact of chemotherapy agents on human primordial follicle reserve. Cancer Res. 2007 Nov 1;67(21):10159-62. doi: 10.1158/0008-5472.CAN-07-2042. PMID 17974956
- [Background] Detti L, Martin DC, Williams RW, Schlabritz-Loutsevich N, Williams LJ, Uhlmann RA. Somatic and reproductive outcomes in mice treated with cyclophosphamide in pre-pubertal age. Syst Biol Reprod Med. 2013 Jun;59(3):140-5. doi: 10.3109/19396368.2012.751463. Epub 2013 Jan 2. PMID 23278118
- [Background] Wallace WH, Thomson AB, Kelsey TW. The radiosensitivity of the human oocyte. Hum Reprod. 2003 Jan;18(1):117-21. doi: 10.1093/humrep/deg016. PMID 12525451
- [Background] Critchley HO, Wallace WH. Impact of cancer treatment on uterine function. J Natl Cancer Inst Monogr. 2005;(34):64-8. doi: 10.1093/jncimonographs/lgi022. PMID 15784827
- [Background] Sarafoglou K, Boulad F, Gillio A, Sklar C. Gonadal function after bone marrow transplantation for acute leukemia during childhood. J Pediatr. 1997 Feb;130(2):210-6. doi: 10.1016/s0022-3476(97)70345-7. PMID 9042122
- [Background] Chemaitilly W, Mertens AC, Mitby P, Whitton J, Stovall M, Yasui Y, Robison LL, Sklar CA. Acute ovarian failure in the childhood cancer survivor study. J Clin Endocrinol Metab. 2006 May;91(5):1723-8. doi: 10.1210/jc.2006-0020. Epub 2006 Feb 21. PMID 16492690
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Kawashima T, Hudson MM, Meadows AT, Friedman DL, Marina N, Hobbie W, Kadan-Lottick NS, Schwartz CL, Leisenring W, Robison LL; Childhood Cancer Survivor Study. Chronic health conditions in adult survivors of childhood cancer. N Engl J Med. 2006 Oct 12;355(15):1572-82. doi: 10.1056/NEJMsa060185. PMID 17035650
- [Background] Green DM, Sklar CA, Boice JD Jr, Mulvihill JJ, Whitton JA, Stovall M, Yasui Y. Ovarian failure and reproductive outcomes after childhood cancer treatment: results from the Childhood Cancer Survivor Study. J Clin Oncol. 2009 May 10;27(14):2374-81. doi: 10.1200/JCO.2008.21.1839. Epub 2009 Apr 13. PMID 19364956
- [Background] Sanchez-Serrano M, Crespo J, Mirabet V, Cobo AC, Escriba MJ, Simon C, Pellicer A. Twins born after transplantation of ovarian cortical tissue and oocyte vitrification. Fertil Steril. 2010 Jan;93(1):268.e11-3. doi: 10.1016/j.fertnstert.2009.09.046. Epub 2009 Oct 31. PMID 19880105
- [Background] Rosendahl M, Schmidt KT, Ernst E, Rasmussen PE, Loft A, Byskov AG, Andersen AN, Andersen CY. Cryopreservation of ovarian tissue for a decade in Denmark: a view of the technique. Reprod Biomed Online. 2011 Feb;22(2):162-71. doi: 10.1016/j.rbmo.2010.10.015. Epub 2010 Nov 16. PMID 21239230
- [Background] Donnez J, Silber S, Andersen CY, Demeestere I, Piver P, Meirow D, Pellicer A, Dolmans MM. Children born after autotransplantation of cryopreserved ovarian tissue. a review of 13 live births. Ann Med. 2011;43(6):437-50. doi: 10.3109/07853890.2010.546807. Epub 2011 Jan 13. PMID 21226660
- [Background] Jeruss JS, Woodruff TK. Preservation of fertility in patients with cancer. N Engl J Med. 2009 Feb 26;360(9):902-11. doi: 10.1056/NEJMra0801454. No abstract available. PMID 19246362
- [Background] Schover LR. Rates of postcancer parenthood. J Clin Oncol. 2009 Jan 20;27(3):321-2. doi: 10.1200/JCO.2008.19.7749. Epub 2008 Dec 15. No abstract available. PMID 19075256
- [Background] Rosen A, Rodriguez-Wallberg KA, Rosenzweig L. Psychosocial distress in young cancer survivors. Semin Oncol Nurs. 2009 Nov;25(4):268-77. doi: 10.1016/j.soncn.2009.08.004. PMID 19879433
- [Background] Byrne J, Fears TR, Steinhorn SC, Mulvihill JJ, Connelly RR, Austin DF, Holmes GF, Holmes FF, Latourette HB, Teta MJ, et al. Marriage and divorce after childhood and adolescent cancer. JAMA. 1989 Nov 17;262(19):2693-9. PMID 2810602
- [Background] Kremer LC, Mulder RL, Oeffinger KC, Bhatia S, Landier W, Levitt G, Constine LS, Wallace WH, Caron HN, Armenian SH, Skinner R, Hudson MM; International Late Effects of Childhood Cancer Guideline Harmonization Group. A worldwide collaboration to harmonize guidelines for the long-term follow-up of childhood and young adult cancer survivors: a report from the International Late Effects of Childhood Cancer Guideline Harmonization Group. Pediatr Blood Cancer. 2013 Apr;60(4):543-9. doi: 10.1002/pbc.24445. Epub 2012 Dec 31. PMID 23281199
- [Background] Oktay K, Karlikaya G. Ovarian function after transplantation of frozen, banked autologous ovarian tissue. N Engl J Med. 2000 Jun 22;342(25):1919. doi: 10.1056/NEJM200006223422516. No abstract available. PMID 10877641
- [Background] Oktay K, Buyuk E, Veeck L, Zaninovic N, Xu K, Takeuchi T, Opsahl M, Rosenwaks Z. Embryo development after heterotopic transplantation of cryopreserved ovarian tissue. Lancet. 2004 Mar 13;363(9412):837-40. doi: 10.1016/S0140-6736(04)15728-0. PMID 15031026
- [Background] Donnez J, Dolmans MM. Cryopreservation and transplantation of ovarian tissue. Clin Obstet Gynecol. 2010 Dec;53(4):787-96. doi: 10.1097/GRF.0b013e3181f97a55. PMID 21048445
- [Background] Donnez J, Jadoul P, Squifflet J, Van Langendonckt A, Donnez O, Van Eyck AS, Marinescu C, Dolmans MM. Ovarian tissue cryopreservation and transplantation in cancer patients. Best Pract Res Clin Obstet Gynaecol. 2010 Feb;24(1):87-100. doi: 10.1016/j.bpobgyn.2009.09.003. Epub 2009 Oct 21. PMID 19850531
- [Background] Silber S, Kagawa N, Kuwayama M, Gosden R. Duration of fertility after fresh and frozen ovary transplantation. Fertil Steril. 2010 Nov;94(6):2191-6. doi: 10.1016/j.fertnstert.2009.12.073. Epub 2010 Feb 19. PMID 20171622
- [Background] Schmidt KL, Byskov AG, Nyboe Andersen A, Muller J, Yding Andersen C. Density and distribution of primordial follicles in single pieces of cortex from 21 patients and in individual pieces of cortex from three entire human ovaries. Hum Reprod. 2003 Jun;18(6):1158-64. doi: 10.1093/humrep/deg246. PMID 12773440
- [Background] Liu J, Van der Elst J, Van den Broecke R, Dhont M. Early massive follicle loss and apoptosis in heterotopically grafted newborn mouse ovaries. Hum Reprod. 2002 Mar;17(3):605-11. doi: 10.1093/humrep/17.3.605. PMID 11870111
- [Background] Gook DA, Edgar DH. Cryopreservation of the human female gamete: current and future issues. Hum Reprod. 1999 Dec;14(12):2938-40. doi: 10.1093/humrep/14.12.2938. No abstract available. PMID 10601074
- [Background] Gook DA, McCully BA, Edgar DH, McBain JC. Development of antral follicles in human cryopreserved ovarian tissue following xenografting. Hum Reprod. 2001 Mar;16(3):417-22. doi: 10.1093/humrep/16.3.417. PMID 11228205
- [Background] Maltaris T, Beckmann MW, Binder H, Mueller A, Hoffmann I, Koelbl H, Dittrich R. The effect of a GnRH agonist on cryopreserved human ovarian grafts in severe combined immunodeficient mice. Reproduction. 2007 Feb;133(2):503-9. doi: 10.1530/REP-06-0061. PMID 17307918
- [Background] Oktem O, Oktay K. The role of extracellular matrix and activin-A in in vitro growth and survival of murine preantral follicles. Reprod Sci. 2007 May;14(4):358-66. doi: 10.1177/1933719107303397. PMID 17644808
- [Background] Soleimani R, Heytens E, Oktay K. Enhancement of neoangiogenesis and follicle survival by sphingosine-1-phosphate in human ovarian tissue xenotransplants. PLoS One. 2011 Apr 29;6(4):e19475. doi: 10.1371/journal.pone.0019475. PMID 21559342
- [Background] Abir R, Fisch B, Jessel S, Felz C, Ben-Haroush A, Orvieto R. Improving posttransplantation survival of human ovarian tissue by treating the host and graft. Fertil Steril. 2011 Mar 15;95(4):1205-10. doi: 10.1016/j.fertnstert.2010.07.1082. PMID 20817170
- [Background] Zelinski MB, Murphy MK, Lawson MS, Jurisicova A, Pau KY, Toscano NP, Jacob DS, Fanton JK, Casper RF, Dertinger SD, Tilly JL. In vivo delivery of FTY720 prevents radiation-induced ovarian failure and infertility in adult female nonhuman primates. Fertil Steril. 2011 Mar 15;95(4):1440-5.e1-7. doi: 10.1016/j.fertnstert.2011.01.012. PMID 21316047
- [Background] Qu J, Godin PA, Nisolle M, Donnez J. Distribution and epidermal growth factor receptor expression of primordial follicles in human ovarian tissue before and after cryopreservation. Hum Reprod. 2000 Feb;15(2):302-10. doi: 10.1093/humrep/15.2.302. PMID 10655299
- [Background] Van den Broecke R, Liu J, Handyside A, Van der Elst JC, Krausz T, Dhont M, Winston RM, Hovatta O. Follicular growth in fresh and cryopreserved human ovarian cortical grafts transplanted to immunodeficient mice. Eur J Obstet Gynecol Reprod Biol. 2001 Aug;97(2):193-201. doi: 10.1016/s0301-2115(00)00507-8. PMID 11451548
- [Background] Keros V, Xella S, Hultenby K, Pettersson K, Sheikhi M, Volpe A, Hreinsson J, Hovatta O. Vitrification versus controlled-rate freezing in cryopreservation of human ovarian tissue. Hum Reprod. 2009 Jul;24(7):1670-83. doi: 10.1093/humrep/dep079. Epub 2009 Apr 9. PMID 19359339
- [Background] Gosden R. Cryopreservation: a cold look at technology for fertility preservation. Fertil Steril. 2011 Aug;96(2):264-8. doi: 10.1016/j.fertnstert.2011.06.029. Epub 2011 Jun 30. PMID 21718989
- [Background] Dolmans MM, Marinescu C, Saussoy P, Van Langendonckt A, Amorim C, Donnez J. Reimplantation of cryopreserved ovarian tissue from patients with acute lymphoblastic leukemia is potentially unsafe. Blood. 2010 Oct 21;116(16):2908-14. doi: 10.1182/blood-2010-01-265751. Epub 2010 Jul 1. PMID 20595517
- [Background] Shaw JM, Bowles J, Koopman P, Wood EC, Trounson AO. Fresh and cryopreserved ovarian tissue samples from donors with lymphoma transmit the cancer to graft recipients. Hum Reprod. 1996 Aug;11(8):1668-73. doi: 10.1093/oxfordjournals.humrep.a019467. PMID 8921114
- [Background] Gosden RG, Rutherford AJ, Norfolk DR. Transmission of malignant cells in ovarian grafts. Hum Reprod. 1997 Mar;12(3):403. doi: 10.1093/humrep/12.3.403. No abstract available. PMID 9130724
- [Background] Rosendahl M, Andersen MT, Ralfkiaer E, Kjeldsen L, Andersen MK, Andersen CY. Evidence of residual disease in cryopreserved ovarian cortex from female patients with leukemia. Fertil Steril. 2010 Nov;94(6):2186-90. doi: 10.1016/j.fertnstert.2009.11.032. Epub 2010 Jan 25. PMID 20100619
- [Background] Moomjy M, Rosenwaks Z. Ovarian tissue cryopreservation: the time is now. Transplantation or in vitro maturation: the time awaits. Fertil Steril. 1998 Jun;69(6):999-1000. doi: 10.1016/s0015-0282(98)00091-0. No abstract available. PMID 9627282
- [Background] Kim SS, Radford J, Harris M, Varley J, Rutherford AJ, Lieberman B, Shalet S, Gosden R. Ovarian tissue harvested from lymphoma patients to preserve fertility may be safe for autotransplantation. Hum Reprod. 2001 Oct;16(10):2056-60. doi: 10.1093/humrep/16.10.2056. PMID 11574491
- [Background] Kauffman HM, McBride MA, Delmonico FL. First report of the United Network for Organ Sharing Transplant Tumor Registry: donors with a history of cancer. Transplantation. 2000 Dec 27;70(12):1747-51. doi: 10.1097/00007890-200012270-00014. PMID 11152107
- [Background] Myron Kauffman H, McBride MA, Cherikh WS, Spain PC, Marks WH, Roza AM. Transplant tumor registry: donor related malignancies. Transplantation. 2002 Aug 15;74(3):358-62. doi: 10.1097/00007890-200208150-00011. PMID 12177614
- [Background] Meirow D, Hardan I, Dor J, Fridman E, Elizur S, Ra'anani H, Slyusarevsky E, Amariglio N, Schiff E, Rechavi G, Nagler A, Ben Yehuda D. Searching for evidence of disease and malignant cell contamination in ovarian tissue stored from hematologic cancer patients. Hum Reprod. 2008 May;23(5):1007-13. doi: 10.1093/humrep/den055. Epub 2008 Mar 15. PMID 18344563
- [Background] Radford JA, Lieberman BA, Brison DR, Smith AR, Critchlow JD, Russell SA, Watson AJ, Clayton JA, Harris M, Gosden RG, Shalet SM. Orthotopic reimplantation of cryopreserved ovarian cortical strips after high-dose chemotherapy for Hodgkin's lymphoma. Lancet. 2001 Apr 14;357(9263):1172-5. doi: 10.1016/s0140-6736(00)04335-x. PMID 11323045
- [Background] Schroder CP, Timmer-Bosscha H, Wijchman JG, de Leij LF, Hollema H, Heineman MJ, de Vries EG. An in vitro model for purging of tumour cells from ovarian tissue. Hum Reprod. 2004 May;19(5):1069-75. doi: 10.1093/humrep/deh244. Epub 2004 Apr 7. PMID 15070872
- [Background] Informed consent, parental permission, and assent in pediatric practice. Committee on Bioethics, American Academy of Pediatrics. Pediatrics. 1995 Feb;95(2):314-7. PMID 7838658
- [Background] Kuther TL. Medical decision-making and minors: issues of consent and assent. Adolescence. 2003 Summer;38(150):343-58. PMID 14560886
- [Background] Gracia CR, Gracia JJ, Chen S. Ethical dilemmas in oncofertility: an exploration of three clinical scenarios. Cancer Treat Res. 2010;156:195-208. doi: 10.1007/978-1-4419-6518-9_15. No abstract available. PMID 20811835